CLINICAL TRIAL: NCT04326491
Title: The Utility of Breath Biopsy as a Screening Tool for HCC: A Pilot Study
Brief Title: The Utility of Breath Biopsy as a Screening Tool for HCC
Acronym: BrtH-C
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 1-085-18
Record Dates: First submitted 2020-03-24; First posted 2020-03-30 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: HCC; Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCC: Participants are diagnosed with HCC on top of cirrhosis
  Interventions: Diagnostic Test: Breath Biopsy
- Cirrhosis with no HCC: Participants are diagnosed with cirrhosis but have no HCC
  Interventions: Diagnostic Test: Breath Biopsy

INTERVENTIONS:
Diagnostic Test: Breath Biopsy — Analysis of breath samples to identify volatile molecules specific to HCC

SUMMARY:
The aim of this pilot study is to examine whether there is a discriminating ability of the breath sample analysis to capture biomarkers specific to the HCC in the breath of affected individuals. If positive, our research could open up a new horizon for cost-effective and feasible screening tools.

DETAILED DESCRIPTION:
20 Participants will be included in the study. Ten Cirrhotic patients with HCC and 10 Cirrhotic patients without HCC.

The first group is patients with HCC secondary to cirrhosis. The second group will be patients with cirrhosis who are currently on the standard surveillance program with no HCC. Confirmation of the absence of HCC would have been ensured via a recent advanced imaging modality (dynamic CT scan or MRI) in the ongoing surveillance programme.

Participants will breathe into either a mouthpiece or collection tube then Breath samples will be analyzed via an analyzer to detect the volatile organic compounds (VOC) and quantitatively compare them

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients with HC.
* Cirrhotic patients without HCC

Exclusion Criteria:

* Patients with more than one primary cancer (HCC in addition to other cancer)
* Patients who are not aware of the diagnosis
* Patients in whom the diagnosis of HCC is not clear and only suspected
* Patients with severe chronic obstructive pulmonary disease (COPD) or severe asthma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is open for participants with liver Cirrhosis (without HCC allocated to an arm) and (with HCC allocated to the other arm). There is no gender restriction.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Volatile organic compounds specific to HCC | 6 months
  Quantitative analysis of the volume and pattern of volatile compounds in the breath of the individuals with HCC compared to that in the breath of individuals without HCC but with the same underlying disease

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Bekheit, PhD, Principal Investigator — NHS Grampian
Locations (1):
- Ashis Mukhopadhya, Aberdeen, United Kingdom